CLINICAL TRIAL: NCT04769505
Title: A Pilot Randomized Controlled Trial to Examine the Feasibility and Effectiveness of a Brief Digital Mindfulness-based Intervention for COPD Patients
Brief Title: Mindfulness-based Interventions in COPD Patients
Acronym: SPIROMIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Landsteiner Institute for Lung Research and Pneumological Oncology (Other)
Collaborators: University of Vienna (Other); Klinik Ottakring (Unknown); Klinik Floridsdorf (Unknown); Therme Wien Med (Ambulant Pulmonary Rehabilitation) (Unknown)
Responsible Party: Principal Investigator, Georg-Christian Funk, Assoc.-Prof. Georg-Christian Funk, M.D., Karl Landsteiner Institute for Lung Research and Pneumological Oncology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPIROMIND 39
Record Dates: First submitted 2021-02-11; First posted 2021-02-24 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants receive a digital mindfulness-based intervention (MBI) + treatment as usual.
  Interventions: Behavioral: digital mindfulness-based intervention (MBI)
- Wait list control group (No Intervention): Participants receive treatment as usual during the intervention period. They are provided with the digital mindfulness-based intervention (MBI) after the intervention period. The waitlist control group receives the same intervention as the intervention group, with the exception of using not using the exercises via the software on the smartphone, but receiving the exercises as audio files.

INTERVENTIONS:
Behavioral: digital mindfulness-based intervention (MBI) — The digital MBI consists of four auditory guided mindfulness exercises lasting between 10 and 15 minutes. The four exercises are a body scan and three sitting meditations (awareness of the heartbeat, awareness of the body, awareness of sounds). The exercises can be conducted via a software (https://www.movisens.com/de/produkte/movisensxs/) on participants' smartphones. Participants will be familiarized with the concept of mindfulness and the intervention in a single face-to-face introductory session. Additionally, participants will receive a manual, containing all relevant information. Participants will be instructed to practice at least once daily over the course of eight weeks. We recommended to come up with a fixed time point for the mindfulness practice to facilitate a routine. They can choose individually between the exercises. After the intervention period, participants received the exercises as audio files and could continue practicing.
  Arms: Intervention group

SUMMARY:
The purpose of this pilot study is to assess the feasibility of a brief digital mindfulness-based intervention for COPD patients and its effectiveness regarding the reduction of psychological distress as well as stress.

DETAILED DESCRIPTION:
Background:

Patients with chronic obstructive pulmonary disease (COPD) do not only suffer from somatic symptoms but also from symptoms of anxiety and depression (defined as psychological distress) as well as stress. As pharmacological interventions showed only limited effectiveness in targeting the latter, a need for additional treatment options emerges. In other chronic conditions, mindfulness-based interventions (MBIs) are effective in reducing symptoms of psychological distress and stress. Despite first promising results, research on MBIs in COPD patients is still scarce and mixed regarding their effects. Furthermore, it is crucial to implement mental health interventions adapted to the needs of COPD patients. Due to often experienced physical limitations and impaired mobility, digital MBIs seem particularly promising.

Aim and Research Questions:

Building on the above, this pilot randomized controlled trial aims to examine a) the feasibility of a brief digital MBI for COPD patients and b) its effects on psychological distress and stress.

Methods:

30 psychologically distressed (assessed by the Hospital Anxiety and Depression Scale, HADS-A ≥ 8 or HADS-D ≥ 8) COPD patients are screened for inclusion and exclusion criteria in a telephone interview and randomly assigned to the MBI (plus treatment as usual) or waitlist control group (treatment as usual). After a single face-to-face introductory session, patients in the MBI condition are instructed to conduct at least one of four brief audio-guided mindfulness exercises (10-15min) daily for 8 weeks, delivered on their smartphones. Following an ecological momentary approach, psychological and respiratory variables (e.g. subjective stress, dyspnoea) are assessed before and after each exercise. These data will be analysed using multilevel modelling. Moreover, primary (psychological distress) and secondary outcomes (e.g. chronic stress, fatigue) are measured at baseline, 4 weeks, 8 weeks, and follow-up, including questionnaires and assessments of biological stress markers (hair cortisol, heart rate variability, electrodermal activity). The data will be analysed using repeated measures ANOVAs. Finally, in semi-structured telephone exit interviews with 15 patients of the MBI group, the intervention's feasibility will be explored using a thematic analysis approach.

ELIGIBILITY:
Inclusion criteria:

1. spirometry confirmed (FEV1<80%) COPD diagnosis
2. psychological distress (as assessed by the Hospital Anxiety and Depression Scale): HADS-A ≥ 8 OR HADS-D ≥ 8 OR*
3. age ≥ 40 years
4. ability to understand German
5. physical and mental capability to attend the intervention, judged by the treating physician
6. life expectancy > 6 months as judged by treating physician
7. ability to use a smartphone
8. ability not to smoke for the duration of the measurement time points (2-3 hours) (This criterion has been added later, because we learned that this was a problem for some participants. However, smoking during the measurements heavily affects biomarker data and the subjective stress response to a stress induction protocol.)

Exclusion Criteria:

1. auditory impairment
2. active asthma diagnosis ("Regardless of your COPD, have you had allergies and asthma in childhood or adolescence and needed medication for them at that time?" If no: No active asthma. If yes: "Is your asthma active and a problem now in addition to your COPD and do you currently need asthma medications because of it?" If no: No active asthma. If yes: exclusion)**
3. any other known severe comorbidities such as heart failure (LVF<35%), uncontrolled diabetes, concomitant cancer, stroke, unstable coronary heart disease, respiratory failure
4. history of/current severe psychological disorder (e.g. schizophrenia, severe cognitive impairment)
5. current acute exacerbation of COPD
6. any other relevant acute health crisis interfering with the study intervention (e.g. Covid-19)
7. receiving any psychosocial treatment (e.g. psychotherapy)
8. regular other systematic mind-body-practice

(*) When the only exclusion criterion was the HADS, which was often the case, we contacted the participants two months later to screen them again and included them, if they were eligible.

(**) We further specified this criterion, as we learned that many patients were told to probably have asthma without them knowing exactly if they had an active asthma diagnosis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Psychological distress | baseline - 4 weeks
  Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983; German version Herrmann-Lingen et al., 2011), scores: 0-42, lower scores indicate improvement, interpreting both subscales for anxiety and depression
Psychological distress | baseline - 8 weeks
  Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983; German version Herrmann-Lingen et al., 2011), scores: 0-42, lower scores indicate improvement, interpreting both subscales for anxiety and depression
Patient's experiences with the digital MBI | 8 weeks
  patients' experiences assessed in the exit interview (qualitative and quantitative data)

SECONDARY OUTCOMES:
Chronic stress | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  assessed by Perceived Stress Scale (PSS-10; Cohen & Williamson, 1988; German version Klein et al., 2016), scores 0-40, lower scores indicate improvement
Health related quality of life | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  Chronic Respiratory Questionnaire (CRQ-SAS; German version Schünemann et al., 2003), scores: 20-140, higher scores indicate improvement
Health status impairment | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  COPD Assessment Test (CAT; Jones et al., 2009), scores 0-40, lower scores indicate improvement
Fatigue | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  Multidimensional Fatigue Inventory (MFI-20; German version Schwarz, Krauss, & Hinz, 2003), scores 0-80, items have different polarity
Mindfulness | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  Freiburger Mindfulness Inventory short form (FMI short form; Walach, Buchheld, Buttenmüller, Kleinknecht, & Schmidt, 2006), scores 0-42, higher scores indicate improvement
Self-compassion | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  Self-Compassion Scale short form (SCS short form; Raes, Pommier, Neff, & Van Gucht, 2011; German version Hupfeld & Ruffieux, 2011), scores 12-60, items have different polarity
Breathlessness catastrophizing | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  Breathlessness Catastrophizing Scale (BCS; Solomon et al., 2015; German version adapted analogue to Pain Catastrophizing Scale Meyer, Sprott, & Mannion, 2008), scores 0-52, lower scores indicate improvement
Stress reactivity | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  the reactivity to stress assessed via examining heart rate variability (RMSSD) during the exposure to a mental stressor (stroop test)
Stress reactivity | baseline, 4 weeks, 8 weeks, 4 months, 6 months
  the reactivity to stress assessed via examining skin conductance level during the exposure to a mental stressor (stroop test)
Hair cortisol | baseline, 8 weeks, 4 months, 6 months
  concentration of hair cortisol (as biomarker for chronic stress)
Psychological distress | baseline, 4 months, 6 months
  Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983; German version Herrmann-Lingen et al., 2011), scores: 0-42, lower scores indicate improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Ottakring, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschenett H, Vafai-Tabrizi F, Zwick RH, Valipour A, Funk GC, Nater UM. Digital mindfulness-based intervention for people with COPD - a multicentre pilot and feasibility RCT. Respir Res. 2025 May 26;26(1):199. doi: 10.1186/s12931-025-03243-4. PMID 40420253

DOCUMENTS (1):
  • Study Protocol (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT04769505/Prot_002.pdf